CLINICAL TRIAL: NCT04790331
Title: Comparative Study Between the Efficacy of Oral Verapamil and Oral Diltiazim on Reduction of Intraoperative Bleeding During Endoscopic Sinus Surgery Under General Anesthesia
Brief Title: Efficacy of Oral Verapamil and Oral Diltiazim on Reduction of Intraoperative Bleeding During Endoscopic Sinus Surgery Under General Anesthesia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Maher Zaki Habeeb, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Verapamil andDiltiazim in ESS
Record Dates: First submitted 2021-02-19; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Verapamil; Diltiazim; FESS
MeSH Terms: interventions — Verapamil; Diltiazem

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- verapamil group (Experimental): verapamil group who will receive verapamil 80 mg PO 3 hours preoperative
  Interventions: Drug: Verapamil
- Ditiazim (Experimental): Diltiazim group will receive Diltiazim 90mg PO 3 hours preoperative
  Interventions: Drug: Diltiazem
- placebo group (Experimental): Placebo oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verapamil — Verapamil is a phenylalkylamine calcium channel blocker used in the treatment of high blood pressure, heart arrhythmias, and angina
  Other Names: Isoptin
  Arms: verapamil group
Drug: Diltiazem — Diltiazem is a calcium channel blocker. It works by relaxing the muscles of your heart and blood vessels.
  Diltiazem is used to treat hypertension and angina.
  Arms: Ditiazim
Drug: Placebo — Placebo oral tablet
  Arms: placebo group

SUMMARY:
To study the effect of addition of oral verapamil or Diltiazim to general anaesthesia on the Intraoperative haemodynamics : heart rate(HR), noninvasive blood pressure(NIBP), mean arterial blood pressure(MAP), and the blood loss during endoscopic sinus surgery.

DETAILED DESCRIPTION:
Functional Endoscopic Sinus Surgery (FESS) is a minimally invasive technique used to restore sinus ventilation and function in patients with recurrent acute or chronic infective sinusitis in whom medical therapy has failed. The term FESS is used to draw attention to the potential for reestablishing natural mucociliary clearance mechanism, drainage and aeration of sinuses, and maintaining as much of the normal anatomy as possible. Over last few years this technique has become popular worldwide due to its minimally invasive nature and preservation of mucosa(1) .

Intraoperative bleeding presents a larger obstacle to endoscopic visualization. Blood obscures the anatomy of the surgical field and dirties the endoscope lens leading to great difficulty in visualization (2). Continued bleeding into the surgical field during FESS not only impairs endoscopic vision , but also can lead to complications including : brain injury, orbital or optic nerve injury, and catastrophic bleeding from major vessels (e.g., internal carotid artery) (2,3).

Endoscopic reconstruction with vascularized tissue is desirable to facilitate rapid healing(4).

Various approaches have been used to secure a dry operating field , among them : conventional anesthesia , total intravenous anesthesia (TIVA) has been previously reported to result in reduced blood loss when used for FESS .

However, few recent studies point out that (TIVA) may not significantly reduce blood loss. (5,6)

One way to achieve this goal "reduction of bleeding" is to induce controlled hypotension For half a century, controlled hypotension has been used to reduce bleeding and need for blood transfusions and provide a satisfactory bloodless surgical field . Controlled hypotension is defined as a reduction of the systolic blood pressure to 80-90mm Hg,a reduction of mean arterial pressure "MAP" to 50-65mmHg or a 30% reduction of baseline "MAP"(7). Pharmacological agents used include those agents , that can be used successfully alone and those that are used adjunctively to limit dosage requirements and therefore , The adverse effects of the other agents . Agents used successfully alone include inhalation anesthetics , sodium Nitroprusside , nitroglycerin , trimethaphon camsilate , alprostadil (prostaglandin E1) , adenosine , remifentanil and agents used in spinal anesthesia.Agents that can be used alone or in combination include :Calcium Channel antagonists ( e.g nicardipine) , beta adrenoceptor - antagonists ( beta-blockers ) e.g bisoprolol , propranolol , esmolol ) and fenoldopam. Agents that are mainly used adjunctively include ACE Inhibitors , and clonidine . The definition of the ideal hypotensive agent is : It must be easy to administer , have a short onset time , an effect that disappears quickly when administration is discontinued , a rapid elimination without toxic metabolites , negligible effects on vital organs and a predictable and dose dependent effect. New agents and techniques have been recently evaluated for their ability to induce effective hypotension without impairing the perfusion of vital organs .(7,8,9)

Calcium channel blockers are drugs that block the entry of calcium into the muscle cells of the heart and arteries. Thus, by blocking the entry of calcium, calcium channel blockers reduce electrical conduction within the heart, decrease the force of contraction (work) of the muscle cells, and dilate arteries which reduces blood pressure and thereby the effort the heart must exert to pump blood(10) .

Although calcium channel blockers have a similar mechanism of action, they differ in their ability to affect heart muscle vs. arteries, and they differ in their ability to affect heart rate and contraction. For example; verapamil (Covera-HS, Verelan PM, Calan , Isoptin) and diltiazim( cardizem , dilacor , tiazac , diltiaxl ), reduces the strength and rate of the heart's contraction and are used in treating abnormal heart rhythms(10

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years.
* patients of both genders.
* ASA grade I - II.

Exclusion Criteria:

* Patient refusal.
* Any contraindication of B- blocker:

  1. Athma , COPD
  2. Bradycardia , Heart block
  3. Acute decompensated heart failure
  4. Peripheral vascular disease
* Any contraindication of calcium channel blocker:

  1. AV conduction defects (2nd and 3rd degree AV block).
  2. Sick sinus syndrome .
  3. Wolf-Parkinson-White Syndrome.
  4. History of congestive heart failure.
  5. Patients on long-term ß-blocker therapy.
  6. Patients with allergy to medication included in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
heart rate | for the duration of surgery up to 2 hours
  heart beats for minutes
Estimated Blood Loss | for the duration of surgery up to 2 hours
  Estimated blood loss in milliliters per hour is calculated by subtracting the volume of total irrigation used during the case from the total amount of fluid in the suction canister at the end of surgery dividing by surgical time in hours.

SECONDARY OUTCOMES:
The Boezaart and van der Merwe intraoperative surgical field scale. | for the duration of surgery up to 2 hours
  Boezaart Bleeding Scale (BBS) (0 - no bleeding (cadaveric conditions), 1 - Slight bleeding, no suctioning required, 2 - Slight bleeding, occasional suctioning required, 3 - Slight bleeding, frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed, 4 - Moderate bleeding, frequent suctioning required, and bleeding threatens surgical field directly after suction is removed, 5 - Severe bleeding, constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible)
plasma norepinephrine concentrations | baseline before anesthesia ( in the holding area with insertion of I.V. cannula) and three hours after the end of surgery.
  plasma norepinephrine concentrations measured by enzyme immunoassay as venous blood samples about 4ml will be collected from each patient under aseptic condition
serum cortisol concentrations | baseline before anesthesia ( in the holding area with insertion of I.V. cannula) and three hours after the end of surgery.
  serum cortisol will be measured by enzyme immunoassay as venous blood samples about 4ml will be collected from each patient under aseptic condition

REFERENCES:
- [Background] Thongrong C, Kasemsiri P, Carrau RL, Bergese SD. Control of bleeding in endoscopic skull base surgery: current concepts to improve hemostasis. ISRN Surg. 2013 Jun 13;2013:191543. doi: 10.1155/2013/191543. Print 2013. PMID 23844295
- [Background] Hadad G, Bassagasteguy L, Carrau RL, Mataza JC, Kassam A, Snyderman CH, Mintz A. A novel reconstructive technique after endoscopic expanded endonasal approaches: vascular pedicle nasoseptal flap. Laryngoscope. 2006 Oct;116(10):1882-6. doi: 10.1097/01.mlg.0000234933.37779.e4. PMID 17003708
- [Background] Stammberger H. Endoscopic endonasal surgery--concepts in treatment of recurring rhinosinusitis. Part II. Surgical technique. Otolaryngol Head Neck Surg. 1986 Feb;94(2):147-56. doi: 10.1177/019459988609400203. PMID 3083327
- [Background] Stankiewicz JA, Lal D, Connor M, Welch K. Complications in endoscopic sinus surgery for chronic rhinosinusitis: a 25-year experience. Laryngoscope. 2011 Dec;121(12):2684-701. doi: 10.1002/lary.21446. Epub 2011 Nov 15. PMID 22086769
- [Background] Eberhart LH, Folz BJ, Wulf H, Geldner G. Intravenous anesthesia provides optimal surgical conditions during microscopic and endoscopic sinus surgery. Laryngoscope. 2003 Aug;113(8):1369-73. doi: 10.1097/00005537-200308000-00019. PMID 12897561
- [Background] Ankichetty SP, Ponniah M, Cherian V, Thomas S, Kumar K, Jeslin L, Jeyasheela K, Malhotra N. Comparison of total intravenous anesthesia using propofol and inhalational anesthesia using isoflurane for controlled hypotension in functional endoscopic sinus surgery. J Anaesthesiol Clin Pharmacol. 2011 Jul;27(3):328-32. doi: 10.4103/0970-9185.83675. PMID 21897501
- [Background] Degoute CS, Ray MJ, Manchon M, Dubreuil C, Banssillon V. Remifentanil and controlled hypotension; comparison with nitroprusside or esmolol during tympanoplasty. Can J Anaesth. 2001 Jan;48(1):20-7. doi: 10.1007/BF03019809. PMID 11212044
- [Background] Tobias JD. Controlled hypotension in children: a critical review of available agents. Paediatr Drugs. 2002;4(7):439-53. doi: 10.2165/00128072-200204070-00003. PMID 12083972
- [Background] Degoute CS. Controlled hypotension: a guide to drug choice. Drugs. 2007;67(7):1053-76. doi: 10.2165/00003495-200767070-00007. PMID 17488147